CLINICAL TRIAL: NCT02424084
Title: Effects of Extracorporeal Shock Wave Therapy in Bone Microcirculation
Brief Title: Bone Microcirculation After Extracorporeal Shock Wave Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Tobias Kisch, MD, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 14-266-4
Record Dates: First submitted 2015-03-31; First posted 2015-04-22 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Intact Scaphoid Bone; Intact Metacarpal Bone; Fractured Scaphoid Bone; Fractured Metacarpal Bone
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Intact scaphoid bone (Experimental): Group A (n=20): Consent-capable male and female patients ≥18 years of age who have an intact scaphoid.
  Intervention: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
  Interventions: Device: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
- Intact metacarpal bone (Experimental): Group B (n=20): Consent-capable male and female patients ≥18 years of age who have an intact metacarpal bone.
  Intervention: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
  Interventions: Device: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
- Fractured scaphoid bone (Experimental): Group C (n=20): Consent-capable male and female patients ≥18 years of age who have a fractured scaphoid.
  Intervention: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
  Interventions: Device: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
- Fractured metacarpal bone (Experimental): Group D (n=20): Consent-capable male and female patients ≥18 years of age who have a fractured metacarpal bone.
  Intervention: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
  Interventions: Device: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
- Intact metatarsal bone (Experimental): Group B (n=20): Consent-capable male and female patients ≥18 years of age who have an intact metatarsal bone.
  Intervention: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)
  Interventions: Device: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave)

INTERVENTIONS:
Device: Extracorporeal Shock Wave Therapy (Device Name: PiezoWave) — Extracorporeal Shock Wave Therapy

SUMMARY:
In trauma surgery and hand surgery treatment strategies of none healing bone fractures aim at replacing pseudarthrosis by well vascularized bone and improving microcirculation. Although previous studies indicate that extracorporeal shock wave therapy (ESWT) can accelerate bone healing in case of non-union, only a few studies focused on the elucidation of its mechanisms of action. Therefore, the aim of this study is to evaluate the microcirculatory effects of extracorporeal shock wave therapy on scaphoid bones and metacarpal and metatarsal in a human in-vivo setting for the first time.

ELIGIBILITY:
Inclusion Criteria:

* Group A (n=20): Consent-capable male and female patients ≥18 years of age who have an intact scaphoid.
* Group B (n=20): Consent-capable male and female patients ≥18 years of age who have an intact metacarpal bone.
* Group C (n=20): Consent-capable male and female patients ≥18 years of age who have a fractured scaphoid.
* Group D (n=20): Consent-capable male and female patients ≥18 years of age who have a fractured metacarpal bone.

Exclusion Criteria:

* below 18 years of age
* scar tissue above scaphoid or metacarpal bone
* osteoporosis or comparable bone disease
* medication that influences bones

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2023-02 (Actual); Study Completion 2023-02 (Actual)

PRIMARY OUTCOMES:
Change in microcirculation (composite outcome measure) | Baseline and 1 minute post-dose
  * Bone blood flow [arbitrary units AU]
  * Bone blood velocity [AU]
  * Tissue oxygen saturation [%]
  * Relative postcapillary venous filling pressure [AU] (Composite outcome measure)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Kisch, MD, Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- University of Schleswig-Holstein, Lübeck, Schleswig-Holstein, Germany